CLINICAL TRIAL: NCT02696148
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Liraglutide in Obese Children Aged 7 to 11 Years
Brief Title: A Trial to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Liraglutide in Obese Children Aged 7 to 11 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-4181; U1111-1162-9171 (Other: WHO); 2014-004454-34 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — For subcutaneous (s.c., under the skin) injection once daily.
  Arms: Liraglutide
Drug: placebo — For subcutaneous (s.c., under the skin) injection once daily.
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America. The aim of this trial is to investigate safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of liraglutide in obese children aged 7 to 11 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 7-11 years (both inclusive) at the time of signing informed consent
* Tanner stage 1 (including subjects with premature adrenarche) at the time of signing informed consent
* BMI (body mass index) corresponding to above or equal to 30 kg/m^2 for adults by international cut-off points (Cole et al 2000)1 and BMI below or equal to 45 kg/m^2 as well as BMI above or equal to 95th percentile for age and gender

Exclusion Criteria:

* Subjects with secondary causes of childhood obesity (i.e., hypothalamic, genetic or endocrine causes)
* Subjects with confirmed bulimia nervosa disorder
* Diagnosis of type 1 diabetes mellitus or type 2 diabetes mellitus as defined by glycosylated haemoglobin (HbA1C) Above or equal to 6.5 %
* History of pancreatitis (acute or chronic)
* Presence of severe co-morbidities as judged by the investigator
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid carcinoma (MTC)
* History of major depressive disorder within 2 years before randomisation

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From the time of first dosing and until completion of follow-up visit (59-108 days after first dosing)

SECONDARY OUTCOMES:
Area under the liraglutide concentration curve | From 0-24 hours at steady state following the last dose (49-91 days after first dosing)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, New Haven, Connecticut
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Pensacola, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Mastrandrea LD, Witten L, Carlsson Petri KC, Hale PM, Hedman HK, Riesenberg RA. Liraglutide effects in a paediatric (7-11 y) population with obesity: A randomized, double-blind, placebo-controlled, short-term trial to assess safety, tolerability, pharmacokinetics, and pharmacodynamics. Pediatr Obes. 2019 May;14(5):e12495. doi: 10.1111/ijpo.12495. Epub 2019 Jan 17. PMID 30653847
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com